CLINICAL TRIAL: NCT00509366
Title: Phase II Prospective Study Evaluating the Role of Personalized Chemotherapy Regimens for Chemo-Naive Select Stage IIIB and IV Non-Small Cell Lung Cancer (NSCLC) in Patients Using a Genomic Predictor of Platinum Resistance to Guide Therapy
Brief Title: Study Using a Genomic Predictor of Platinum Resistance to Guide Therapy in Stage IIIB/IV Non-Small Cell Lung Cancer
Acronym: TOP0602
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to reproducibility issues with genomics prediction model.
Sponsor: Duke University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004599
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: genomics; genomics predictor; genomics analysis; squamous; non-squamous
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cisplatin Sensitive (Post-Amendment) (Active Comparator): Assignment to Treatment Group based on histology and tumor genomics analysis:
  Squamous Cell NSCLC-Cisplatin day 1, Gemcitabine days 1 & 8 Non-Squamous Cell NSCLC-Cisplatin day 1, Pemetrexed day 1
  Per an amendment dated 1/25/2010, post-amendment treatment assignment refers to the further separation of patients into sub-groups, within the cisplatin sensitive arm, based on histology (squamous/non-squamous).
  Interventions: Drug: Cisplatin & Gemcitabine; Drug: Cisplatin & Pemetrexed
- Cisplatin Resistant (Post-Amendment) (Active Comparator): Assignment to Treatment Group based on histology and tumor genomics analysis:
  Squamous Cell NSCLC-Docetaxel day 1, Gemcitabine days 1 & 8 Non-Squamous Cell NSCLC-Pemetrexed day 1, Gemcitabine days 1 & 8
  Per an amendment dated 1/25/2010, post-amendment treatment assignment refers to the further separation of patients into sub-groups, within the cisplatin resistant arm, based on histology (squamous/non-squamous).
  Interventions: Drug: Docetaxel & Gemcitabine; Drug: Pemetrexed & Gemcitabine
- Cisplatin Sensitive (Pre-Amendment) (Active Comparator): Assignment to Treatment Group based on tumor genomics analysis:
  Cisplatin day 1, Gemcitabine days 1 & 8
  Interventions: Drug: Cisplatin & Gemcitabine
- Cisplatin Resistant (Pre-Amendment) (Active Comparator): Assignment to Treatment Group based on tumor genomics analysis:
  Pemetrexed day 1, Gemcitabine days 1 & 8
  Interventions: Drug: Pemetrexed & Gemcitabine

INTERVENTIONS:
Drug: Cisplatin & Gemcitabine — Squamous Cell NSCLC:
  Gemcitabine 1250 mg/m2 IV over 30 minutes day 1 and 8, followed by Cisplatin 75 mg/m2 IV over 60 minutes day 1; repeat every 21 days for up to 6 cycles
  Other Names: Gemzar
  Arms: Cisplatin Sensitive (Post-Amendment); Cisplatin Sensitive (Pre-Amendment)
Drug: Cisplatin & Pemetrexed — Non-Squamous Cell NSCLC:
  Pemetrexed 500 mg/m2 IV over approximately 10 minutes day 1, followed by Cisplatin 75 mg/m2 IV over 60 minutes day 1; repeat every 21 days for up to 6 cycles
  Other Names: Alimta
  Arms: Cisplatin Sensitive (Post-Amendment)
Drug: Docetaxel & Gemcitabine — Squamous Cell NSCLC:
  Docetaxel 75 mg/m2 IV over 60 minutes day 1, followed by Gemcitabine 1250 mg/m2 IV over 30-60 minutes day 1 and alone day 8; repeat every 21 days for up to 6 cycles
  Other Names: Taxotere; Gemzar
  Arms: Cisplatin Resistant (Post-Amendment)
Drug: Pemetrexed & Gemcitabine — Non-Squamous Cell NSCLC:
  Pemetrexed 500 mg/m2 IV over approximately 10 minutes day 1, followed by Gemcitabine 1250 mg/m2 IV over 30-60 minutes day 1 and alone day 8; repeat every 21 days for up to 6 cycles
  Other Names: Alimta; Gemzar
  Arms: Cisplatin Resistant (Post-Amendment); Cisplatin Resistant (Pre-Amendment)

SUMMARY:
In this trial, subjects with chemo-naive advanced non-small cell lung cancer (NSCLC) were assigned to chemotherapy using a genomic-based predictor for platinum sensitivity. After an amendment dated 1/25/2010, subjects with squamous cell NSCLC sensitive to cisplatin received cisplatin/gemcitabine and if resistant to cisplatin received docetaxel/gemcitabine. Subjects with non-squamous cell NSCLC sensitive to cisplatin received cisplatin/pemetrexed and if resistant to cisplatin received pemetrexed/gemcitabine. The primary objective of this trial was to prospectively validate the genomic-based prediction model through separate evaluation of the one-year progression-free survival (PFS) of the cisplatin-sensitive and cisplatin-resistant cohorts. Secondary objectives included: assessment of overall time to progressive disease, quality of life and evaluation of drug sensitivity patterns of cisplatin and pemetrexed.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in both men and women. The majority of patients with lung cancer have non-small cell type (NSCLC). The current standard of care for treating select stage IIIB and stage IV NSCLC is a doublet chemotherapy regimen, such as cisplatin plus gemcitabine, carboplatin plus paclitaxel, or a platinum agent plus vinorelbine. All of these regimens have comparable response rates as first-line therapy. In addition, the combination of cisplatin plus pemetrexed has recently been approved for non-squamous histology, based on results of a large randomized prospective trial in advanced stage NSCLC. Alternative doublet therapy for first-line treatment of NSCLC per ASCO and NCCN guidelines also include a non-platinum doublet or single agent therapy.

An individual patient's response to chemotherapy is the result of complex interactions between the drug(s) and the patient's genetics and environment. Using Affymetrix gene expression data with corresponding drug response data for cisplatin from the NCI60 lines panel, a gene expression based model predicative of cisplatin-resistant has been developed. However, reevaluation of the genomics-based prediction model showed that it was irreproducible, suggesting inaccurate patient assignments into the two cisplatin cohorts. As a result, it would be inappropriate to separately analyze outcomes for the different treatment groups. Instead, information from both cisplatin cohorts will be combined to reflect the overall measure of one-year progression-free survival in this study. Secondary outcomes will also reflect the overall measures of median time to disease progression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or histologic/cytologic select stage IIIB or IV NSCLC, not amenable to curative treatment with surgery or XRT. Histologic/cytologic documentation of recurrence required in patients who were previously completely resected and now have metastatic disease.
* Fresh frozen tissue must be available to generate and apply the genomics predictor. If not obtained at the time of diagnosis, then subject must consent to another biopsy as a fresh tissue sample must yield adequate high quality RNA. Patients with symptomatic brain metastases must complete brain XRT and be neurologically stable (steroids permitted) prior to research biopsy. If patient had prior XRT therapy, fresh frozen tissue biopsy for genomics analysis must be outside XRT field.
* At least one, non-radiated, measurable lesion by RECIST criteria.
* ECOG performance status of 0 or 1.
* NO prior chemo, biologic or targeted therapy for any malignancy. Prior therapy with low dose methotrexate or similar medications allowed if used for non-malignant conditions.
* Prior XRT therapy is permitted if ≥1 week since completion of XRT (≥2 weeks for whole brain XRT). XRT must be <25% of bone marrow reserve.
* Age ≥18 years.
* No previous or concomitant malignancy in past 5 years other than surgical management for carcinoma in situ of the cervix, breast, NSCLC, basal cell or squamous cell carcinoma of the skin.
* No other serious medical or psychiatric illness.
* Signed informed consent.
* Required lab data within 2 weeks of enrollment:

  1. ANC/AGC ≥1500 per uL
  2. Platelets ≥100,000 per uL
  3. Total bili ≤1.5 mg/dL
  4. Creatinine ≤2 mg/dL; creatinine clearance ≥45 ml/min.
  5. SGOT/SGPT ≤3x ULN except in presence of known hepatic mets (may be up to 5x ULN) unless receive docetaxel/gemcitabine than SGOT/SGPT ≤1.5x ULN.
* Females of child-bearing potential (not surgically sterilized and between menarche and 1 year post menopause) must test negative for pregnancy within 7 days prior to or at the time of enrollment based on a serum pregnancy test.
* Both sexually active males and females of reproductive potential must agree to use a reliable method of birth control, as determine by the patient and their health care team, during study and for 3 months following the last dose of study drug.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Concurrent administration of any other anti-tumor therapy (see #5 inclusion for exceptions).
* Inability to comply with protocol or study procedures.
* Active infection requiring IV antibiotics, antifungal or antiviral agents, that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Untreated CNS metastases unless brain XRT completed and neurologically stable (steroids permitted).
* Major surgery within 2 weeks of study or other serious concomitant systemic disorders that would compromise the safety of the patient or patient's ability to complete the study.
* MI having occurred less than 6 months before inclusion, any known uncontrolled arrhythmia, symptomatic angina pectoris, active ischemia or cardiac failure not controlled by meds.
* Contraindications to corticosteroids.
* Inability/unwillingness to take folic acid or vitamin B12.
* Unwillingness to stop taking herbal supplements while on study.
* Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to treatment initiation and throughout study enrollment.
* Inability to discontinue aspirin at a dose >1300 mg/day or other non-steroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days for long-acting agents such as piroxicam).
* Female patients that are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Vlahovic, MD, MHS, Principal Investigator — Duke University
Locations (8):
- United States (8):
  - Duke University Medical Center, Durham, North Carolina
  - Maria Parham Hospital, Henderson, North Carolina
  - Scotland HealthCare System (Scotland Memorial Hospital), Laurinburg, North Carolina
  - Southeastern Regional Medical Center, Gibson Cancer Center, Lumberton, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Coastal Cancer Center, Myrtle Beach, South Carolina
  - Community Memorial Health Center, South Hill, Virginia

REFERENCES:
- [Background] Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Genomic signatures to guide the use of chemotherapeutics. Nat Med. 2006 Nov;12(11):1294-300. doi: 10.1038/nm1491. Epub 2006 Oct 22. PMID 17057710 (Retraction: PMID 21217686 Potti A, Dressman HK, Bild A, Riedel RF, Chan G, Sayer R, Cragun J, Cottrill H, Kelley MJ, Petersen R, Harpole D, Marks J, Berchuck A, Ginsburg GS, Febbo P, Lancaster J, Nevins JR. Nat Med. 2011 Jan;17(1):135)
- [Background] Bild AH, Yao G, Chang JT, Wang Q, Potti A, Chasse D, Joshi MB, Harpole D, Lancaster JM, Berchuck A, Olson JA Jr, Marks JR, Dressman HK, West M, Nevins JR. Oncogenic pathway signatures in human cancers as a guide to targeted therapies. Nature. 2006 Jan 19;439(7074):353-7. doi: 10.1038/nature04296. Epub 2005 Nov 6. PMID 16273092
- See also: Clinical Trials at Duke Comprehensive Cancer Center — http://www.cancer.duke.edu/CTrials/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin + Gemcitabine: Cisplatin Sensitive patients were registered at the start of the study and assigned to cisplatin + gemcitabine protocol-based treatment consistent with histology. One patient who was assigned to this arm withdrew from the study. This patient did not receive protocol treatment and was classified as a screen failure.
- Cisplatin + Pemetrexed: Cisplatin Sensitive patients were registered at the start of the study and assigned to cisplatin + pemetrexed protocol-based treatment consistent with histology. One patient who was assigned to this arm was deemed ineligible due to the discover of brain metastasis. This patient did not receive protocol treatment and was classified as a screen failure.
- Pemetrexed + Gemcitabine: Cisplatin Resistant patients were registered at the start of the study and assigned to pemetrexed + gemcitabine protocol-based treatment consistent with histology. One patient who was assigned to this arm was later deemed ineligible before initiating protocol treatment and was classified as a screen failure.
- Docetaxel + Gemcitabine: Cisplatin Resistant patients were registered at the start of the study and assigned to docetaxel+ gemcitabine protocol-based treatment consistent with histology.
- Screen Failure: Screen failures constitute patients who were registered into the study but were not assigned to treatment due to unsuccessful genomic analysis. Nine patients did not undergo biopsy. Eight experienced complications from biopsy. The remaining 34 were deemed ineligible after genomic screening. Note that three patients who were assigned protocol-based treatment (2 in the cisplatin sensitive group and 1 in the cisplatin resistant group) did not receive the treatment and were added to the 51 initially identified as screen failures within the summary of baseline characteristics and outcome measures.
Period: Overall Study
Arm/Group | Cisplatin + Gemcitabine | Cisplatin + Pemetrexed | Pemetrexed + Gemcitabine | Docetaxel + Gemcitabine | Screen Failure
Started | 18 (Registered patients who were assigned cisplatin/gemcitabine treatment.) | 8 (Registered patients who were assigned cisplatin/pemetrexed treatment.) | 22 (Registered patients who were assigned pemetrexed/gemcitabine treatment.) | 2 (Registered patients who were assigned docetaxel/gemcitabine treatment.) | 51 (Registered patients who were neither assigned nor treated with protocol-based therapy.)
Assigned Treatment | 18 (Patients who were assigned to cisplatin/gemcitabine treatment arm.) | 8 (Patients who were assigned to cisplatin/pemetrexed treatment arm.) | 22 (Patients who were assigned to pemetrexed/gemcitabine treatment arm.) | 2 (Patients who were assigned to docetaxel/gemcitabine treatment arm.) | 0
Completed | 17 (Patients assigned to treatment and treated with cisplatin/gemcitabine treatment combination.) | 7 (Patients assigned to treatment and treated with cisplatin/pemetrexed treatment combination.) | 21 (Patients assigned to treatment and treated with pemetrexed/gemcitabine treatment combination.) | 2 (Patients assigned to treatment and treated with docetaxel/gemcitabine treatment combination.) | 51 (Patients who were neither assigned nor treated with protocol-based therapy.)
Not Completed | 1 | 1 | 1 | 0 | 0
Not completed — Not Treated (Screen Failure) | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants in each group reflects the number of participants at the end of the study period (COMPLETED) in the Participant Flow Analysis, with the exception of 3 patients who were assigned treatment, but not treated, and were added to the number of screen failures.
Groups:
- Cisplatin + Gemcitabine: Cisplatin Sensitive patients were registered at the start of the study, assigned to cisplatin/gemcitabine protocol-based treatment consistent with histology, and treated during the course of the study.
- Cisplatin + Pemetrexed: Cisplatin Sensitive patients were registered at the start of the study, assigned to cisplatin/pemetrexed protocol-based treatment consistent with histology, and treated during the course of the study.
- Pemetrexed + Gemcitabine: Cisplatin Resistant patients were registered at the start of the study, assigned to cisplatin/gemcitabine resistant protocol-based treatment consistent with histology, and treated during the course of the study.
- Docetaxel + Gemcitabine: Cisplatin Resistant patients were registered at the start of the study, assigned to docetaxel/gemcitabine resistant protocol-based treatment consistent with histology, and treated during the course of the study.
- Screen Failure: Screen failures constitute patients who were registered into the study but were not assigned to treatment due to unsuccessful genomic analysis or those who were assigned treatment but not treated after reevaluation of their eligibility.
- Total: Total of all reporting groups
Arm/Group | Cisplatin + Gemcitabine | Cisplatin + Pemetrexed | Pemetrexed + Gemcitabine | Docetaxel + Gemcitabine | Screen Failure | Total
Number analyzed (Participants) | 17 | 7 | 21 | 2 | 54 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.53 (6.51) | 61.43 (9.78) | 62.14 (9.72) | 59.00 (7.07) | 61.24 (10.10) | 61.61 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 9 | 0 | 20 | 40
  Male | 11 | 2 | 12 | 2 | 34 | 61
Region of Enrollment [Number; unit: participants]
  United States | 17 | 7 | 21 | 2 | 54 | 101

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression Free Survival Rate in Chemo-naive Select Stage IIIB or Stage IV NSCLC Patients
Description: One-year progression-free survival was defined from the time from initiation of study treatment to the first date of disease progression or death as a result of any cause. Progression was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Time was censored at the date of the last follow-up visit for patients who were still alive and have not progressed. The one-year progression free survival rate is a percentage, representing the fraction of treated patients who, after one-year, are disease free or alive.
Time Frame: 1 year
Population: Due to the irreproducible nature of the genomic signatures of cisplatin sensitivity, analyses based on separate treatment groups were inappropriate. Therefore, all enrolled participants (initiated for treatment) from both treatment arms were analyzed together.
Measure: Number (95% Confidence Interval); unit: percentage of treated patients
Groups:
- Treatment: Treatment refers to the combined cisplatin sensitive and resistant arms of the study. Due to the irreproducibility of the genomics-based prediction model for assigning patients into the original cisplatin treatment arms, patients from both arms were combined for analysis.
Arm/Group | Treatment
Number analyzed (Participants) | 47
percentage of treated patients | 19.15 [9.46 to 31.40]

2. Secondary Outcome: Median Time to Progressive Disease
Description: Median time to progressive disease was defined as the time from enrollment to the the time at which 50% of patients had experienced disease progression. Enrollment is defined as having successful genomic analysis and start of chemotherapy. Time was censored at date of death for patients who have not had documented disease progression, at first available date of other anti-tumor therapy for patients who were either administered other anti-tumor therapy prior to documented disease progression or administered other anti-tumor therapy without documented disease progression, and at last date of followup if neither non-protocol therapy was administered nor progression documented.
Time Frame: 1 Year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 47
months | 4.60 [3.58 to 6.47]

3. Secondary Outcome: Mean Change From Baseline to Follow-up Cycle in Quality of Life - Functional Assessment of Cancer Therapy-Lung (FACT-L)
Description: The outcome measure is mean change in the Trial Outcome Index (TOI) between baseline and each follow-up assessment measured by the Functional Assessment of Cancer Therapy-Lung (FACT-L). The FACT-L instrument consists of 34 items to assess physical (PWB), social and family (SWB), emotional (EWB), functional well-being (FWB) and additional lung specific concerns (LCS). Using a 5-point Likert type scale, responses to individual items range from 0 (not at all) to 4 (Very Much) with higher scores indicating better quality of life. The TOI is the sum of PWB (7 items), FWB (7 items) and LCS scores (7 items), which each have a possible range between 0 and 28. Therefore, TOI ranges from 0 to 84.
Time Frame: Baseline, Every 21 days for a maximum of 6 cycles
Population: Of the 50 patients assigned treatment, only 32 patients completed the FACT-L assessment at baseline and at least one follow-up.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Treatment: Treatment refers to the combined cisplatin sensitive (cisplatin/pemetrexed or cisplatin/gemcitabine) and resistant (pemetrexed/gemcitabine or docetaxel/gemcitabine) arms of the study. Due to the irreproducibility of the genomics-based prediction model for assigning patients into the original cisplatin treatment arms, patients from both arms were combined for analysis.
Arm/Group | Treatment
Number analyzed (Participants) | 32
units on a scale
  Change from baseline to Cycle 1 | 0.15 (1.76)
  Change from baseline to Cycle 2 | -1.04 (2.23)
  Change from baseline to Cycle 3 | -1.28 (2.97)
  Change from baseline to Cycle 4 | -2.62 (2.48)
  Change from baseline to Cycle 5 | -6.14 (3.96)
  Change from baseline to Cycle 6 | -0.72 (3.20)

4. Secondary Outcome: Drug Sensitivity Quartiles for Cisplatin and Pemetrexed
Description: Using genomics-based prediction models previously developed separately for cisplatin and pemetrexed, the probability that each patient was sensitive or would respond to treatment was computed. Quartiles describe the patterns of drug sensitivity probabilities. The 1st, 2nd, and 3rd quartiles are the sensitivity levels at which 25%, 50%, and 75% of patients have lower sensitivity.
Time Frame: 3 years
Population: This outcome is not summarized due to irreproducibility of the genomics-based prediction model and resulting probability estimates.
Groups:
- Treatment: Treatment refers to the combined cisplatin sensitive and resistant arms of the study.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: May 2007 to December 2011
Groups:
- Cisplatin Sensitive (Pre-Amendment): Pre-amendment cisplatin sensitive refers to patients who experienced adverse events and treated with cisplatin-sensitive protocol based therapy per the amendment dated 1/25/2010.
- Cisplatin Sensitive (Post-Amendment): Post-amendment cisplatin sensitive refers to patients who experienced adverse events and treated with cisplatin-sensitive protocol based therapy per the amendment dated AFTER 1/25/2010.
- Cisplatin Resistant (Pre-Amendment): Pre-amendment cisplatin resistant refers to patients who experienced adverse events and treated with cisplatin-resistant protocol based therapy per the amendment dated 1/25/2010.
- Cisplatin Resistant (Post-Amendment): Pre-amendment cisplatin sensitive refers to patients who experienced adverse events and treated with cisplatin-sensitive protocol based therapy per the amendment dated AFTER 1/25/2010.
- Screen Failure: Screen failures constitute patients who were registered into the study and underwent protocol-based procedure (e.g. biopsy, genomic screening), but were not enrolled to genomics-directed, protocol-based therapy. From the participant flow, 9 of the 54 screen failures did not have adverse event follow-up, resulting in a final count of 45 screen failures with adverse event follow-up.
Arm/Group | Cisplatin Sensitive (Pre-Amendment) | Cisplatin Sensitive (Post-Amendment) | Cisplatin Resistant (Pre-Amendment) | Cisplatin Resistant (Post-Amendment) | Screen Failure
Serious Adverse Events (participants affected / at risk) | 8/16 | 5/8 | 12/17 | 4/6 | 3/45
Other Adverse Events (participants affected / at risk) | 16/16 | 8/8 | 17/17 | 6/6 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin Sensitive (Pre-Amendment) (N=16) | Cisplatin Sensitive (Post-Amendment) (N=8) | Cisplatin Resistant (Pre-Amendment) (N=17) | Cisplatin Resistant (Post-Amendment) (N=6) | Screen Failure (N=45)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Asystole (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 2 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0
Infections and infestations - Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Vagina (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin Sensitive (Pre-Amendment) (N=16) | Cisplatin Sensitive (Post-Amendment) (N=8) | Cisplatin Resistant (Pre-Amendment) (N=17) | Cisplatin Resistant (Post-Amendment) (N=6) | Screen Failure (N=45)
Anemia (Blood and lymphatic system disorders) | 14 | 6 | 15 | 6 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 3 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 3 | 1 | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 7 | 3 | 0 | 0 | 0
Blurred vision (Eye disorders) | 3 | 0 | 4 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 2 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye disorders - Other (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Flashing lights (Eye disorders) | 0 | 0 | 1 | 0 | 0
Watering eyes (Eye disorders) | 1 | 0 | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 7 | 12 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 2 | 6 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 2 | 6 | 3 | 0
Nausea (Gastrointestinal disorders) | 13 | 8 | 12 | 2 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 6 | 4 | 0 | 0
Chills (General disorders) | 3 | 2 | 4 | 2 | 0
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 7 | 2 | 10 | 2 | 0
Edema trunk (General disorders) | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 13 | 7 | 15 | 5 | 0
Fever (General disorders) | 3 | 3 | 9 | 4 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 2 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Immune system disorders - Other (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gum infection (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Infections and infestations-Infection with Grade 3 or 4 neutrophils: Skin (cellulitis) (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2 | 14 | 4 | 0
Alkaline phosphatase increased (Investigations) | 7 | 4 | 11 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 10 | 5 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 0
Creatinine increased (Investigations) | 9 | 4 | 2 | 1 | 0
Investigations - Other (Investigations) | 1 | 4 | 2 | 2 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 11 | 4 | 12 | 6 | 0
Platelet count decreased (Investigations) | 9 | 5 | 8 | 4 | 0
Weight gain (Investigations) | 2 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 4 | 2 | 4 | 3 | 0
White blood cell decreased (Investigations) | 9 | 3 | 12 | 6 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 12 | 5 | 9 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 2 | 2 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 6 | 14 | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 5 | 14 | 6 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 5 | 11 | 4 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 10 | 5 | 5 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 4 | 2 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 10 | 5 | 9 | 6 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 1 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 11 | 3 | 7 | 2 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 2 | 6 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Olfactory nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 9 | 0 | 5 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 3 | 4 | 3 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 6 | 4 | 3 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 3 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 11 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 5 | 8 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 2 | 11 | 3 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The microarray-based prediction model of chemotherapy sensitivity, used to allocate patients into the cisplatin treatment arms, was irreproducible and inaccurate. Quality of life measurements were incomplete and could not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No